CLINICAL TRIAL: NCT00596999
Title: A Single-Arm Study to Assess the Safety of Transplantation With Umbilical Cord Blood Augmented With Human Placental-Derived Stem Cells From Partially Matched Related Donors in Subjects With Certain Malignant Hematologic Diseases and Non-Malignant Disorders
Brief Title: A Single-arm Safety Study of Transplantation Using Umbilical Cord Blood and Human Placental-derived Stem Cells From Partially Matched Related Donors in Persons With Certain Malignant Blood Diseases and Non-malignant Disorders
Acronym: HPDSC
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Organization: Celgene (Industry)
Other Study IDs: CCT-HPDSC-001
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2007-11

CONDITIONS: Hematologic Malignancies
Keywords: Myelodysplastic Syndrome (MDS); Acute myelogenous Leukemia (AML); Acute Lymphocytic Leukemia (ALL); Sickle Cell Disease (SCD); Beta Thalassemia; Inborn Errors of Metabolism; Severe Combined Immunodeficiency Disease (SCID)
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Sickle Cell; beta-Thalassemia; Metabolism, Inborn Errors; X-Linked Combined Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: all subjects will be treated with UCB and HPDSC
  Interventions: Procedure: UCB and HPDSC

INTERVENTIONS:
Procedure: UCB and HPDSC — single dose of UCB followed by one unit of HPDSC

SUMMARY:
To investigate the safety of partially matched related human placental-derived stem cells (HPDSC) administered in conjunction with umbilical cord blood (UCB) stem cells from the same donor in subjects with various malignant or nonmalignant disorders potentially curable with stem cell transplantation and to assess potential restoration of normal hematopoiesis and immune function in subjects with these disorders

ELIGIBILITY:
Inclusion Criteria:

* suitable UCB collected from partially or fully HLA matched related donor
* subject requires umbilical cord transplantation

Exclusion Criteria:

* any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* major anticipated illness or organ failure incompatible with survival from stem cell transplant

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: subjects requiring cord blood transplantation
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2007-05; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of GVHD, time to engraftment and survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lolie Yu, MD, Principal Investigator — Louisiana State University Children's Hospital
Locations (1):
- Louisiana State University Children's Hospital, New Orleans, Louisiana, United States